CLINICAL TRIAL: NCT04172558
Title: Intracavernous Injection of Onabotulinumtoxin-A 100 U For Treatment of Phosphodiesterase Type 5 Inhibitors-Inconvenient Patients With Erectile Dysfunction: A Randamized Controlled Trial.
Brief Title: Intracavernous Injection of Botox 100 U for Treatment of PDE5Is Inconvenient Patients With ED
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDIRB2017122601-34
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Erectile Dysfunction
Keywords: Botulimium Toxin; Eractile Dysfunction; ICI
MeSH Terms: conditions — Erectile Dysfunction | interventions — Botulinum Toxins, Type A; trimix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BTX100 group (Active Comparator): ICI of Botox 100 U
  Interventions: Biological: OnabotulinumtoxinA
- Trimix group (Active Comparator): ICI of Trimix
  Interventions: Drug: Trimix

INTERVENTIONS:
Biological: OnabotulinumtoxinA — a single ICI of BTX-A 100 units one day after the penile Doppler/trimix test.
  Other Names: Grroup 1
  Arms: BTX100 group
Drug: Trimix — on demand ICI of Trimix
  Other Names: Group 2
  Arms: Trimix group

SUMMARY:
There is a new emerging concept that Botulinum Toxin Type A may have a potential role in treatment of erectile dysfunction with a longer duration of action. So, the investigators opted to perform this study to compare ICI of Botulinum Toxin Type A versus Trimix for treatment of ED.

DETAILED DESCRIPTION:
Background: Direct Intracavernosal injections of vasoactive agents to treat erectile dysfunction were first described in 1982 using papaverine. Later on many agents have been introduced for ICI. one of most newly introduced ICI agents for treatment of ED is Botulinum Toxin Type A.

Purpose: The aim of this study will to compare the safety, efficacy, tolerability and adverse events s of ICI of BTX-A 100 unit in comparison with ICI Trimix in the treatment of Erectile Dysfunction for PDE5Is non-responders.

Design, Settings, and Participants: This study will be conducted on 124 patients at minimum, complain of erectile dysfunction not responding to different PDE5Is therapy presenting to Urology department and outpatient clinic at Banha University Hospital.

patients will be randomized into 2 equal groups: The treatment group A: will receive a single ICI of BTX-A 100 units . The treatment group B: will receive on-demand ICI of Trimix .

Assessment for all groups will be done by Sexual Health Inventory for men (SHIM), Sexual Encounter Profile questions 2 and 3 (SEP 2 & SEP 3), and the global assessment question (GAQ) based on pre-treatment, 2 weeks, 3 months and every 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 40 years with ED not responding to PDE5Is, non compliant or contraindicated to PDE5Is. A "No" response on Sexual encounter profile questions (SEP 2 & 3)

Exclusion Criteria:

* psychiatric condition Any presence of penile anatomical abnormalities (e.g. penile fibrosis) that would significantly impair erectile function.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 124 (Estimated)
Dates: Start 2019-03-10 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) | baseline, 2 weeks post treatment then every 3 months post treatment
  Changes in the Erectile Function (EF) domain score of the International Index of change of Erectile Function measured by (IIEF) between treatment periods and baseline in the 2 study arms. It ranges between 0 to 25
Dopller study | baseline, 2 weeks post treatment then every 3 months post treatment
  measurement of Cavernosal artery peak systolic and end diastolic velocities before and after ICI
Erection hardness score [ Time Frame: 2 weeks ] [ Designated as safety issue: No ] Clinical assessment of the Erection hardness score by the investigators in both Erection hardness score | baseline, 2 weeks post treatment then every 3 months post treatment
  Erection hardness score which is ranged 0 to 4

SECONDARY OUTCOMES:
Sexual Encounter Profile 2&3 | baseline, 2 weeks post treatment then every 3 months post treatment
  Assessment of SEP before and after ICI. patient answer ' Yes' or 'No'.
Global Assessment Questionnaire | baseline, 2 weeks post treatment then every 3 months post treatment
  Global Assessment Questionnaire with Yes/No response

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Shaer, MD, Principal Investigator — Banha Univesity hosptals
Locations (1):
- Banha University Hospitals, Banhā, Kalubiaya, Egypt